CLINICAL TRIAL: NCT00079963
Title: Gender, Obesity, C-Reactive Protein, and Oxidative Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: University of California, Berkeley (Other); Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 62378DK; R01DK062378 (NIH)
Record Dates: First submitted 2004-03-18; First posted 2004-03-22 (Estimated); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Ascorbic Acid; Vitamin E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- X (Experimental): Vitamin C
  Interventions: Dietary Supplement: Vitamin C
- Y (Experimental): Vitamin E
  Interventions: Dietary Supplement: Vitamin E
- Z (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin C — 1000 mg/day
  Arms: X
Dietary Supplement: Vitamin E — 800 IU/day
  Arms: Y
Dietary Supplement: Placebo
  Arms: Z

SUMMARY:
This randomized placebo-controlled trial will test whether supplementing with vitamins C and E can lower markers of inflammation and oxidative stress in healthy adults. We will examine whether one antioxidant vitamin is more effective than another, and whether gender or body fat influence the treatment effects. We will also determine whether gender, body fat, or menopausal status are associated with baseline concentrations of inflammation and oxidative stress markers.

DETAILED DESCRIPTION:
Participants will be given 1000 mg vitamin C or 800 IU vitamin E daily for 60 days.

ELIGIBILITY:
Inclusion criteria:

* Nonsmoker and not passively exposed
* Males and females 18 year and older
* Able to take vitamin supplements
* Able to take acetominophen instead of aspirin or NSAIDs during the study

Exclusion criteria:

* Pregnancy or lactation
* History of ever smoking or passive smoke exposure in the last year
* Active liver disease; history of HIV/AIDS, diabetes, kidney stones, hemochromatosis, or autoimmune diseases; heart disease, stroke, or cancer in the last 5 years
* User of prescribed anti-inflammatory or lipid-lowering medications, oral contraceptives, hormone replacement therapy, or blood-thinning drugs
* User of iron supplements or vitamin E at 600 IU per day or more
* Consumption of more than 2 alcoholic beverages per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2004-04; Primary Completion 2008-03-24 (Actual); Study Completion 2008-03-24 (Actual)

PRIMARY OUTCOMES:
Change in high-sensitivity C-reactive protein (hsCRP) | 8-week intervention

SECONDARY OUTCOMES:
Change in blood pressure | 8-week intervention
Change in self-reported stress and psychosocial factors | 8-week intervention
Change in oxidative stress biomarkers (F2-Isoprostanes, malondialdehyde) | 8-week intervention
Association of gender, body fat, menopausal status with baseline concentrations of inflammation and oxidative stress biomarkers. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Gladys Block, Ph.D., Principal Investigator — University of California at Berkeley
Locations (1):
- University of California, Berkeley School of Public Health, Berkeley, California, United States

REFERENCES:
- [Result] Block G, Jensen CD, Morrow JD, Holland N, Norkus EP, Milne GL, Hudes M, Dalvi TB, Crawford PB, Fung EB, Schumacher L, Harmatz P. The effect of vitamins C and E on biomarkers of oxidative stress depends on baseline level. Free Radic Biol Med. 2008 Aug 15;45(4):377-84. doi: 10.1016/j.freeradbiomed.2008.04.005. Epub 2008 Apr 16. PMID 18455517
- [Derived] Block G, Shaikh N, Jensen CD, Volberg V, Holland N. Serum vitamin C and other biomarkers differ by genotype of phase 2 enzyme genes GSTM1 and GSTT1. Am J Clin Nutr. 2011 Sep;94(3):929-37. doi: 10.3945/ajcn.111.011460. Epub 2011 Aug 3. PMID 21813807